CLINICAL TRIAL: NCT01561586
Title: Randomized Phase III Clinical Trial of Weekly Versus Tri-weekly Cisplatin Based Chemoradiation in Locally Advanced Cervical Cancer
Brief Title: Tri-weekly Cisplatin Based Chemoradiation in Locally Advanced Cervical Cancer
Acronym: TACO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea Cancer Center Hospital (Other)
Collaborators: Seoul National University Hospital (Other); Asan Medical Center (Other); Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sang-Young Ryu, Chair of Cerivcal/Ovarian Cancer Center, Korea Cancer Center Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KGOG 1027/THAI 2012
Record Dates: First submitted 2012-03-20; First posted 2012-03-23 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Concurrent chemoradiation; Cisplatin
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Weekly cisplatin with RT (Active Comparator): Weekly cisplatin 40mg/m2 six cycles concurrent to radiation therapy
  Interventions: Drug: Weekly cisplatin with RT
- B: Tri-weekly cisplatin with RT (Experimental): Tri-weekly cisplatin 75mg/m2 three cycles concurrent to radiation therapy
  Interventions: Drug: Tri-weekly cisplatin with RT

INTERVENTIONS:
Drug: Weekly cisplatin with RT — Cisplatin 40mg/m2 IV Weekly For 6 Cycles.(The 6th cycle of cisplatin may be omitted if external beam radiation therapy has been completed) Cisplatin may be diluted and administered per established institutional guidelines. For general suggestion, 40 mg/ m2 of cisplatin may be diluted in 250 ml 0.9% sodium chloride and administered over one or two hours.
  Cisplatin will be given on the first day of external RT (Day 1), preferably, and must be given prior to radiation treatment on that day
  External beam RT will be followed by intracavitary brachytherapy. The total elapsed time for completion of external beam to the whole pelvis, intracavitary BT, and parametrial / nodal RT shall not exceed eight weeks (56 days)
  Other Names: Cisplatin
  Arms: A: Weekly cisplatin with RT
Drug: Tri-weekly cisplatin with RT — Tri-weekly cisplatin 75mg/m2 three cycles concurrent to radiation therapy
  Cisplatin may be diluted and administered per established institutional guidelines. For general suggestion, 75 mg/m2 of cisplatin may be diluted in 500 ml 0.9% sodium chloride and administered over one or two hours (rate of 1 mg of cisplatin per minute).
  Cisplatin will be given on the first day of external RT (Day 1), preferably, and must be given prior to radiation treatment on that day.
  External beam RT will be followed by intracavitary brachytherapy. The total elapsed time for completion of external beam to the whole pelvis, intracavitary BT, and parametrial / nodal RT shall not exceed eight weeks (56 days)
  Other Names: Cisplatin
  Arms: B: Tri-weekly cisplatin with RT

SUMMARY:
Current standard treatment for locally advanced cervical cancer is cisplatin-based concurrent chemoradiation (CRT). Although recently reported meta-analysis studies also demonstrated improved local control rates and survival with cisplatin-based chemotherapy concurrent to radiation therapy (RT), the optimal cisplatin dose and dosing schedule are still undetermined.

In light of the results of the previous clinical trial, weekly cisplatin 40 mg/m2 considered to be a standard regiment in cisplatin doses and dosing schedules. However, our randomized phase II trial showed that tri-weekly cisplatin 75mg/m2 has lower toxicities and a better outcome in locally advanced cervical cancer.

In this randomized phase III trial, the investigators investigate that there may be a survival difference between weekly cisplatin 40 mg/m2 and tri-weekly cisplatin 75 mg/m2 administration concurrent to RT in cervical cancer.

DETAILED DESCRIPTION:
Cervical carcinoma is one of the most common gynecologic cancers worldwide. The prognosis of cervical cancer is favorable, with around 80-90% 5-year survival rate in early stage disease. However, advanced disease carries a poor prognosis. Current standard treatment for locally advanced cervical cancer, which is not eligible for surgical treatment, is cisplatin-based concurrent chemoradiation (CRT). Based on the results of five randomized clinical trials, which consistently showed improved survival in patients treated with cisplatin-based CRT, the National Cancer Institute (NCI) of the United States announced that 'Strong consideration should be given to the incorporation of concurrent cisplatin-based chemotherapy with RT in women who require radiation therapy for treatment of cervical cancer' in 1999.

Although recently reported meta-analysis studies also demonstrated improved local control rates and survival with cisplatin-based chemotherapy concurrent to radiation therapy (RT), the optimal cisplatin dose and dosing schedule are still undetermined. Among the previous five randomized clinical trials, two trials performed by the Gynecologic Oncology Group (GOG) used weekly cisplatin 40 mg/m2 while the other three trials used tri-weekly cisplatin at a dosage range of 50 mg/m2 to 75 mg/m2 combined with 5-fluorouracil (5-FU). Despite the diversity in cisplatin dose and dosing schedules, weekly cisplatin at a dose of 40 mg/m2 concurrent to RT is widely accepted as the standard regimen of CRT because of its convenience, equal effectiveness, and favorable toxicity in comparison to other 5-FU combined regimens.

However, as a result of the GOG 165 study, which was closed prematurely because an interim analysis found that patients in the 5-FU treatment group were not likely to achieve a better outcome, the role of 5-FU (previously popularly included in clinical trials) as a radiosensitizer became subject to debate. Furthermore, a clinical trial performed by the NCI in Canada comparing pelvic RT alone with weekly cisplatin 40 mg/m2 concurrent to RT failed to show improvement of progression free and 5-year survival. While the authors suggested several possible reasons for why their study failed to demonstrate a survival benefit with concurrent weekly cisplatin 40 mg/m2 chemotherapy, other investigators have tried to find another optimal dose and dosing schedule for cisplatin administration.

In light of the results of the previous clinical trial that indicated 5-FU may not be an active radiosensitizer, weekly cisplatin 40 mg/m2 and tri-weekly cisplatin 75 mg/m2 remain the most popular cisplatin doses and dosing schedules. However, despite the possible advantages of tri-weekly cisplatin 75 mg/m2, which offer an increased peak concentration of cisplatin and cisplatin administration during brachytherapy, no clinical trials thus far have directly compared weekly and tri-weekly cisplatin-based chemotherapy concurrent to RT.

Recently the investigators reported a randomized phase II trial to compare the compliance to and toxicity of weekly cisplatin 40 mg/m2 and tri-weekly cisplatin 75 mg/m2 administration concurrent to RT. The study showed that tri-weekly cisplatin 75 mg/m2 concurrent to RT is feasible and increase 5-year survival rate significantly compared to weekly cisplatin 40 mg/m2 in patients with locally advanced cervical cancer (66.5% in the weekly arm, 88.7% in the tri-weekly arm; HR=0.375, 95% CI: 0.154-0.914, p= .03).

Therefore, in this randomized phase III trial, The investigators intend to confirm the survival difference between weekly cisplatin 40 mg/m2 and tri-weekly cisplatin 75 mg/m2 administration concurrent to RT in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will have pathologically proven primary locally advanced cervical cancer with squamous cell carcinoma, adenosquamous carcinoma or adenocarcinoma histology suitable for primary treatment with chemoradiation with curative intent
* FIGO 2008 stage 1B2, 2B, 3B, 4A
* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have adequate Hematologic function(ANC ≥ 1,500/mcl and platelets ≥ 100,000/mcl), Renal function(serum creatinine ≤ ULN or calculated creatinine clearance ≥ 60 mL/min), Hepatic function(serum bilirubin ≤ 1.5 x ULN and AST ≤ 2.5 x ULN and ALT≤ 2.5 x ULN)
* Patients must have signed an approved informed consent

Exclusion Criteria:

* Patients with cervix cancer who have received any previous radiation or chemotherapy
* Patients assessed at presentation as requiring interstitial brachytherapy treatment
* FIGO stage 3A disease
* Para-aortic nodal involvement above the level of the common iliac nodes or L3/L4 (if biopsy proven, PET positive or > 15mm short axis diameter on CT)
* Patients with bilateral hydronephrosis unless at least one side has been stented and renal function fulfils the required inclusion criteria
* Previous chemotherapy for this tumor
* Evidence of distant metastases
* Prior diagnosis of Crohn's disease or ulcerative colitis
* Patients who are pregnant or lactating
* History of other invasive malignancies, with the exception of non-melanoma skin cancer and in situ melanoma, who had (or have) any evidence of the other cancer present within the last 5 years
* Serious illness or medical condition that precludes the safe administration of the trial treatment including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2012-03 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From entry into the study to 5 year after treatment or death
  Observed length of life from entry into the study to death; or for living patients, the date of last contact regardless of whether or not this contact is on a subsequent protocol.

SECONDARY OUTCOMES:
Progression Free Survival | 5 year after treatment
  The time from randomization to the time of disease progression as determined by the investigator (by clinical, radiological or pathological means) or death from any cause
Recurrence rate | 5 year after therapy
  Clinical, radiological or histological reoccurrence of disease since study entry.
  Site of First Recurrence (e.g. para-aortic or supraclavicular lymph nodes, lung, liver, bone, etc.) will also be documented.
Adverse events | 5 years after therapy
  Adverse event is any untoward medical occurrence in a patient or clinical investigational subject administered a study treatment and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An adverse event is any adverse change (developing or worsening) from the patient's pre-treatment condition, including intercurrent illness.
Compliance to radiation protocol | 56~ 67 days after treatment start
  Variation acceptable:
  * Total treatment completed within 56 days (+20% = 67 days)
  * Total dose received to Point A inclusive of EBRT and BT = 80 - 86.4 Gy +/- 5%
  Deviation unacceptable:
  * Total treatment greater than 67 days
  * Total dose received at Point A less than 76 Gy or greater than 90.7 Gy

CONTACTS AND LOCATIONS:
Overall Officials: SANG YOUNG SY RYU, M.D., Principal Investigator — STAFF; SARIKAPAN WILAILAK, M.D., Principal Investigator — Ramathibodi Hospital
Locations (15):
- Fudan University Shanghai Cancer Center, Shanghai, China
- South Korea (12):
  - Dongnam Inst.of Radiological/Medical Science, Busan
  - Soon Chun Hyang University Hospital, Cheonan
  - Dongsan Medical Center, Daegu
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Gachon University Gil Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea Cancer Center Hospital, Korea Institute of Radiological & Medical Sciences, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyungpook National University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital/Sinchon Severance Hospital, Seoul
- Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand
- Ho Chi Minh City Oncology Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Garcia AA, Blessing JA, Darcy KM, Lenz HJ, Zhang W, Hannigan E, Moore DH. Phase II clinical trial of capecitabine in the treatment of advanced, persistent or recurrent squamous cell carcinoma of the cervix with translational research: a gynecologic oncology group study. Gynecol Oncol. 2007 Mar;104(3):572-9. doi: 10.1016/j.ygyno.2006.09.002. Epub 2006 Oct 17. PMID 17049588
- [Background] Keys HM, Bundy BN, Stehman FB, Muderspach LI, Chafe WE, Suggs CL 3rd, Walker JL, Gersell D. Cisplatin, radiation, and adjuvant hysterectomy compared with radiation and adjuvant hysterectomy for bulky stage IB cervical carcinoma. N Engl J Med. 1999 Apr 15;340(15):1154-61. doi: 10.1056/NEJM199904153401503. PMID 10202166
- [Background] Morris M, Eifel PJ, Lu J, Grigsby PW, Levenback C, Stevens RE, Rotman M, Gershenson DM, Mutch DG. Pelvic radiation with concurrent chemotherapy compared with pelvic and para-aortic radiation for high-risk cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1137-43. doi: 10.1056/NEJM199904153401501. PMID 10202164
- [Background] Peters WA 3rd, Liu PY, Barrett RJ 2nd, Stock RJ, Monk BJ, Berek JS, Souhami L, Grigsby P, Gordon W Jr, Alberts DS. Concurrent chemotherapy and pelvic radiation therapy compared with pelvic radiation therapy alone as adjuvant therapy after radical surgery in high-risk early-stage cancer of the cervix. J Clin Oncol. 2000 Apr;18(8):1606-13. doi: 10.1200/JCO.2000.18.8.1606. PMID 10764420
- [Background] Rose PG, Bundy BN, Watkins EB, Thigpen JT, Deppe G, Maiman MA, Clarke-Pearson DL, Insalaco S. Concurrent cisplatin-based radiotherapy and chemotherapy for locally advanced cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1144-53. doi: 10.1056/NEJM199904153401502. PMID 10202165
- [Background] Whitney CW, Sause W, Bundy BN, Malfetano JH, Hannigan EV, Fowler WC Jr, Clarke-Pearson DL, Liao SY. Randomized comparison of fluorouracil plus cisplatin versus hydroxyurea as an adjunct to radiation therapy in stage IIB-IVA carcinoma of the cervix with negative para-aortic lymph nodes: a Gynecologic Oncology Group and Southwest Oncology Group study. J Clin Oncol. 1999 May;17(5):1339-48. doi: 10.1200/JCO.1999.17.5.1339. PMID 10334517
- [Background] Green JA, Kirwan JM, Tierney JF, Symonds P, Fresco L, Collingwood M, Williams CJ. Survival and recurrence after concomitant chemotherapy and radiotherapy for cancer of the uterine cervix: a systematic review and meta-analysis. Lancet. 2001 Sep 8;358(9284):781-6. doi: 10.1016/S0140-6736(01)05965-7. PMID 11564482
- [Background] Chemoradiotherapy for Cervical Cancer Meta-Analysis Collaboration. Reducing uncertainties about the effects of chemoradiotherapy for cervical cancer: a systematic review and meta-analysis of individual patient data from 18 randomized trials. J Clin Oncol. 2008 Dec 10;26(35):5802-12. doi: 10.1200/JCO.2008.16.4368. Epub 2008 Nov 10. PMID 19001332
- [Background] Kirwan JM, Symonds P, Green JA, Tierney J, Collingwood M, Williams CJ. A systematic review of acute and late toxicity of concomitant chemoradiation for cervical cancer. Radiother Oncol. 2003 Sep;68(3):217-26. doi: 10.1016/s0167-8140(03)00197-x. PMID 13129628
- [Background] Lanciano R, Calkins A, Bundy BN, Parham G, Lucci JA 3rd, Moore DH, Monk BJ, O'Connor DM. Randomized comparison of weekly cisplatin or protracted venous infusion of fluorouracil in combination with pelvic radiation in advanced cervix cancer: a gynecologic oncology group study. J Clin Oncol. 2005 Nov 20;23(33):8289-95. doi: 10.1200/JCO.2004.00.0497. Epub 2005 Oct 17. PMID 16230678
- [Background] Pearcey R, Brundage M, Drouin P, Jeffrey J, Johnston D, Lukka H, MacLean G, Souhami L, Stuart G, Tu D. Phase III trial comparing radical radiotherapy with and without cisplatin chemotherapy in patients with advanced squamous cell cancer of the cervix. J Clin Oncol. 2002 Feb 15;20(4):966-72. doi: 10.1200/JCO.2002.20.4.966. PMID 11844818
- [Background] Ryu SY, Lee WM, Kim K, Park SI, Kim BJ, Kim MH, Choi SC, Cho CK, Nam BH, Lee ED. Randomized clinical trial of weekly vs. triweekly cisplatin-based chemotherapy concurrent with radiotherapy in the treatment of locally advanced cervical cancer. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e577-81. doi: 10.1016/j.ijrobp.2011.05.002. Epub 2011 Aug 11. PMID 21840137
- [Background] Mitsuhashi A, Uno T, Tanaka N, Suzuka K, Tate S, Yamazawa K, Matsui H, Yamamoto S, Ito H, Sekiya S. Phase I study of daily cisplatin and concurrent radiotherapy in patients with cervical carcinoma. Gynecol Oncol. 2005 Jan;96(1):194-7. doi: 10.1016/j.ygyno.2004.09.038. PMID 15589600
- [Background] Watanabe Y, Nakai H, Shimaoka M, Tobiume T, Tsuji I, Hoshiai H. Feasibility of concurrent cisplatin use during primary and adjuvant chemoradiation therapy: a phase I study in Japanese patients with cancer of the uterine cervix. Int J Clin Oncol. 2006 Aug;11(4):309-13. doi: 10.1007/s10147-006-0567-4. PMID 16937305
- [Background] Bonomi P, Blessing JA, Stehman FB, DiSaia PJ, Walton L, Major FJ. Randomized trial of three cisplatin dose schedules in squamous-cell carcinoma of the cervix: a Gynecologic Oncology Group study. J Clin Oncol. 1985 Aug;3(8):1079-85. doi: 10.1200/JCO.1985.3.8.1079. PMID 3894589
- [Background] Thigpen T, Shingleton H, Homesley H, LaGasse L, Blessing J. cis-Dichlorodiammineplatinum(II) in the treatment of gynecologic malignancies: phase II trials by the Gynecologic Oncology Group. Cancer Treat Rep. 1979 Sep-Oct;63(9-10):1549-55. PMID 498154
- [Background] Ikushima H, Osaki K, Furutani S, Yamashita K, Kawanaka T, Kishida Y, Iwamoto S, Takegawa Y, Kudoh T, Nishitani H. Chemoradiation therapy for cervical cancer: toxicity of concurrent weekly cisplatin. Radiat Med. 2006 Feb;24(2):115-21. doi: 10.1007/BF02493277. PMID 16715672
- [Background] Chumworathayi B, Suprasert P, Charoenkwan K, Srisomboon J, Phongnarisorn C, Siriaree S, Cheewakriangkrai C, Tantipalakorn J, Kiatpeerakul C, Pantusart A. Weekly versus three-weekly cisplatin as an adjunct to radiation therapy in high-risk stage I-IIA cervical cancer after surgery: a randomized comparison of treatment compliance. J Med Assoc Thai. 2005 Nov;88(11):1483-92. PMID 16471090
- [Background] Monk BJ, Huang HQ, Cella D, Long HJ 3rd; Gynecologic Oncology Group Study. Quality of life outcomes from a randomized phase III trial of cisplatin with or without topotecan in advanced carcinoma of the cervix: a Gynecologic Oncology Group Study. J Clin Oncol. 2005 Jul 20;23(21):4617-25. doi: 10.1200/JCO.2005.10.522. Epub 2005 May 23. PMID 15911864
- [Background] Quasthoff S, Hartung HP. Chemotherapy-induced peripheral neuropathy. J Neurol. 2002 Jan;249(1):9-17. doi: 10.1007/pl00007853. PMID 11954874
- [Background] Maduro JH, Pras E, Willemse PH, de Vries EG. Acute and long-term toxicity following radiotherapy alone or in combination with chemotherapy for locally advanced cervical cancer. Cancer Treat Rev. 2003 Dec;29(6):471-88. doi: 10.1016/s0305-7372(03)00117-8. PMID 14585258
- [Background] Siegal T, Haim N. Cisplatin-induced peripheral neuropathy. Frequent off-therapy deterioration, demyelinating syndromes, and muscle cramps. Cancer. 1990 Sep 15;66(6):1117-23. doi: 10.1002/1097-0142(19900915)66:63.0.co;2-o. PMID 2169332
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Huang HQ, Brady MF, Cella D, Fleming G. Validation and reduction of FACT/GOG-Ntx subscale for platinum/paclitaxel-induced neurologic symptoms: a gynecologic oncology group study. Int J Gynecol Cancer. 2007 Mar-Apr;17(2):387-93. doi: 10.1111/j.1525-1438.2007.00794.x. PMID 17362317
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] McQuellon RP, Thaler HT, Cella D, Moore DH. Quality of life (QOL) outcomes from a randomized trial of cisplatin versus cisplatin plus paclitaxel in advanced cervical cancer: a Gynecologic Oncology Group study. Gynecol Oncol. 2006 May;101(2):296-304. doi: 10.1016/j.ygyno.2005.10.039. Epub 2006 Jan 10. PMID 16376417
- [Background] Cella DF, Wiklund I, Shumaker SA, Aaronson NK. Integrating health-related quality of life into cross-national clinical trials. Qual Life Res. 1993 Dec;2(6):433-40. doi: 10.1007/BF00422217. PMID 8161977
- [Background] Bonomi AE, Cella DF, Hahn EA, Bjordal K, Sperner-Unterweger B, Gangeri L, Bergman B, Willems-Groot J, Hanquet P, Zittoun R. Multilingual translation of the Functional Assessment of Cancer Therapy (FACT) quality of life measurement system. Qual Life Res. 1996 Jun;5(3):309-20. doi: 10.1007/BF00433915. PMID 8763799
- [Background] Eremenco SL, Cella D, Arnold BJ. A comprehensive method for the translation and cross-cultural validation of health status questionnaires. Eval Health Prof. 2005 Jun;28(2):212-32. doi: 10.1177/0163278705275342. PMID 15851774
- [Background] Yun YH, Mendoza TR, Heo DS, Yoo T, Heo BY, Park HA, Shin HC, Wang XS, Cleeland CS. Development of a cancer pain assessment tool in Korea: a validation study of a Korean version of the brief pain inventory. Oncology. 2004;66(6):439-44. doi: 10.1159/000079497. PMID 15452372
- [Background] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- [Background] Cantor AB, Shuster JJ. Parametric versus non-parametric methods for estimating cure rates based on censored survival data. Stat Med. 1992 May;11(7):931-7. doi: 10.1002/sim.4780110710. PMID 1604072
- [Background] Cantor A. Extending SAS Survival Analysis Techniques for Medical Research. Vol. 103. SAS Institute Inc. Cary, NC; 1997.
- [Background] Schoenfeld DA, Richter JR. Nomograms for calculating the number of patients needed for a clinical trial with survival as an endpoint. Biometrics. 1982 Mar;38(1):163-70. PMID 7082758
- [Background] Cantor AB. Sample size calculations for the log rank test: a Gompertz model approach. J Clin Epidemiol. 1992 Oct;45(10):1131-6. doi: 10.1016/0895-4356(92)90153-e. PMID 1474409
- [Background] Lachin JM. Statistical considerations in the intent-to-treat principle. Control Clin Trials. 2000 Jun;21(3):167-89. doi: 10.1016/s0197-2456(00)00046-5. PMID 10822117
- [Background] Agresti A. A survey of exact inference for contingency tables. Statistical Science. 1992; 7: 131-177.
- [Background] Lan KKG., DeMets DL. Discrete sequential boundaries for clinical trials. Biometrika. 1983;70:659-663
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341